CLINICAL TRIAL: NCT00582166
Title: Ibritumomab Tiuxetan Plus Rituximab as Initial Therapy for Patients With High Tumor Burden, Indolent Histology Non-Hodgkin's Lymphoma
Brief Title: Ibritumomab Tiuxetan (Zevalin)+ Rituximab Maintenance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See 'Limitations and Caveats' section
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO04405; NCI-2011-00579 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2018-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Zevalin, High Tumor Burden Indolent Non-Hodgkin's Lymphoma, Ibritumomab Tiuxetan
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibritumomab Tiuxetan (Zevalin) with Rituximab maintenance (Experimental)
  Interventions: Drug: Ibritumomab Tiuxetan (Zevalin) + Rituximab

INTERVENTIONS:
Drug: Ibritumomab Tiuxetan (Zevalin) + Rituximab — Subjects will receive the Ibritumomab Tiuxetan (Zevalin) therapeutic regimen; then rituximab consolidation and maintenance therapy every 3 months until disease progression
  Other Names: Zevalin; Ibritumomab Tiuxetan; Rituximab

SUMMARY:
Subjects will receive the Ibritumomab Tiuxetan (Zevalin) therapeutic regimen; then rituximab consolidation and maintenance therapy every 3 months until disease progression

DETAILED DESCRIPTION:
The objective of this study is to estimate the median progression-free survival for patients receiving this regimen, along with the rate of complete response at 6 months, toxicities associated with this regimen, and laboratory correlates. Subjects will receive the Ibritumomab Tiuxetan (Zevalin) therapeutic regimen; then rituximab consolidation and maintenance therapy every 3 months until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven non-hodgkins lymphoma of follicular grade 1, 2, or 3
* Meeting FLIPI criteria for intermediate or high risk.
* No prior chemotherapy, radiotherapy or immunotherapy for lymphoma;
* Patients may not have known HIV infection, and must not be Hepatitis B Surface Antigen positive.

Exclusion Criteria:

* May not be pregnant or breastfeeding, have documented CNS (Central Nervous System) disease, G-CSF (Granulocyte Colony Stimulating Facto) or GM-CSF (Granulocyte/Macrophage Colony Stimulating Factor) within 2 weeks prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-01-25 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University Of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zevalin With Rituximab Maintenance: Zevalin (Ibritumomab Tiuxetan )+ Rituximab: Subjects will receive the Zevalin(Ibritumomab Tiuxetan) therapeutic regimen; then rituximab consolidation and maintenance therapy every 3 months until disease progression
Period: Overall Study
Arm/Group | Zevalin With Rituximab Maintenance
Started | 18
Completed | 16
Not Completed | 2
Not completed — Death | 1
Not completed — Ineligible pathology | 1

BASELINE CHARACTERISTICS:
Population: Participants with biopsy-proven diagnosis of non-Hodgkin's lymphoma with follicular grade 1, 2, and 3.
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 55 [37 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Estimate median progression free survival (PFS), where PFS is defined as the number of days from administration of Ibritumomab tiuxetan In111 (defined as day 1) until the participant develops progressive disease or death from NHL (Non-Hodgkin's Lymphoma).
Time Frame: up to 5 years, 9.5 months, from first day on treatment to last follow up
Population: The study was stopped prematurely, subjects were not followed for a full 7 years. We have data for 16 subjects, 6 experienced a progression event, 10 survived progression-free through last follow-up. Date of last follow-up is used to calculate progression-free survival for those who did not experience progression.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 16
months | 44.3 [32.8 to 46.1]

2. Secondary Outcome: 24-month Progression Free Survival (PFS)
Description: Estimate the 24 month progression free survival (PFS), where PFS is defined as the number of days from the first Ibritumomab tiuxetan administration (day 0) to the day the patient experiences an event of disease progression (or death). PFS is summarized as the percentage of patients that survived progression free after 24 months.
  Progression is defined as any of the following:
  - Appearances of any new lesions/sites during or after therapy.
  * Increase of >/= 50% in the SPD (sum of perpendicular diameter) from nadir measurement of all involved dominant lymph nodes and liver nodules and spleen nodules or unequivocal progression in any nonmeasurable disease or nondominant site.
  * Increase by > 50% in greatest diameter from nadir measurement of any previously involved dominant node > 1.0 cm in its short axis.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 16
Participants | 11

3. Secondary Outcome: Response Rates
Description: To estimate the Complete Response and unconfirmed Complete Response rate (assessing Ibritumomab tiuxetan). Complete response is defined as the complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related B-symptoms, and all dominant lymph nodes and nodal masses have regressed to normal size, and complete resolution of lymphoma in the bone marrow biopsy. Unconfirmed Complete Response (CRu) defined as the above, but with either a > 1.5cm residual node that has decreased by >75%, and/or individual nodes that were previously confluent that have decreased by >75% in SPD, and/or indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia).
Time Frame: Up to 5 years and 9.5 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 16
percentage of participants | 44 [23 to 67]

4. Secondary Outcome: Number of Participants Experiencing Toxicities, Measured by CTCAE v3.0
Description: To record the toxicities associated with this regimen.
Time Frame: Up to 5 years and 9.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 16
Participants | 16

5. Secondary Outcome: Overall Survival (OS)
Description: To estimate overall survival, 95% confidence intervals will be used.
Time Frame: At 12 months
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zevalin With Rituximab Maintenance
Number analyzed (Participants) | 16
percentage of participants | 93 [80 to 100]

ADVERSE EVENTS:
Arm/Group | Zevalin With Rituximab Maintenance
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin With Rituximab Maintenance (N=16)
Infection (Infections and infestations) | 1 (1) — Infection with grade 3 or 4 neutropenia
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Tranfusion: Platelets (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin With Rituximab Maintenance (N=16)
Auditory/Ear - Other - Vertigo (Ear and labyrinth disorders) | 1 (1)
Blood/Bone Marrow - Other - Anemia (Blood and lymphatic system disorders) | 9 (9)
Leukocytes (Blood and lymphatic system disorders) | 15 (28)
Lymphopenia (Blood and lymphatic system disorders) | 9 (37)
Neutrophils/granulo-cytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (9)
Platelets (Blood and lymphatic system disorders) | 13 (31)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (19)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 109/L (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Dermatology/Skin - Other - Cold Sore (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatology/Skin - Other - Knee Puncture (Skin and subcutaneous tissue disorders) | 1 (1) — Subject indicated involvement in a deer attack
Dermatology/Skin - Other - Rash (erythema & scaling) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other - Skin (Skin and subcutaneous tissue disorders) | 2 (2) — No other information was provided in the study chart other than "Skin"
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Hot Flashes/flushes (Endocrine disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomitting (Gastrointestinal disorders) | 2 (2)
Hemmorage/Bleeding - Other - Hemmorage (Vascular disorders) | 1 (1)
Infection - Dermatology/Skin - Skin (cellulitus) (Infections and infestations) | 1 (1)
Infection - Other - Infection (Infections and infestations) | 3 (5)
Infection - Pulmonary/Upper Respiratory - Sinus (Infections and infestations) | 1 (1)
Infection - Pulmonary/Upper Respiratory - Upper aerodigestive NOS (Infections and infestations) | 1 (3) — "THRUSH" was documented for all events
Infection - Pulmonary/Upper Respiratory - Upper Airway NOS (Infections and infestations) | 4 (5) — "INFECTION - URI [Upper Respiratory Infection]" was documented in all cases
Infection with normal ANC or Grade 1 or 2 neutropenia - Bronchitis (Infections and infestations) | 1 (1)
Edema:limb (Blood and lymphatic system disorders) | 1 (2)
ALT, SGOT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) — ALT (aspartate aminotranferase increased) documented
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other - (PT(INR)) (Metabolism and nutrition disorders) | 1 (1) — INR (international normalized ratio) noted on chart
Metabolic/Laboratory - Other (Sodium - low) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration - anxiety (Psychiatric disorders) | 1 (2)
Neurology - Other - Neuralgia (Nervous system disorders) | 1 (2)
Neurology - Other - Neuro-Sensory (Nervous system disorders) | 1 (3)
Ocular/Vision - Other - Vision Problems (Eye disorders) | 1 (1)
Ocular/Vision - Other - Worsening Peripheral Vision (Eye disorders) | 1 (2)
Pain - Gastrointestinal - Abdomen (Gastrointestinal disorders) | 2 (3)
Pain - Musculoskeletal - Extremity/Limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Musculoskeletal - Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Gastrointestinal - Joint (Musculoskeletal and connective tissue disorders) | 2 (2) — Subject 2 - hip Subject 4 - wrist
Pain - Neurology - Head/Headache (Nervous system disorders) | 4 (4)
Pain - Other - Other (Nervous system disorders) | 3 (3) — Only "PAIN" documented
Pain - Other - Splenamalgy (Immune system disorders) | 1 (1)
Pain - Pulmonary/Upper Respiratory - Pleura (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - Sexual/Reproductive Function - Pelvis (Reproductive system and breast disorders) | 1 (1)
Pain - Musculoskeletal - Muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Gastrointestinal - Tooth (Gastrointestinal disorders) | 2 (2)
Pain - Hepatobiliary/Pancreas - gallbladder (Hepatobiliary disorders) | 1 (1)
Pain - Ocular - Eye (Eye disorders) | 1 (1)
Pain - Other - Groin (Reproductive system and breast disorders) | 1 (1)
Pain - Other - Epigastric (Gastrointestinal disorders) | 1 (1)
Pain - Pulmonary/Upper Respiratory - Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other - Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/genitourinary - Other (Dysuria) (Renal and urinary disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
From IRB: Subjects have completed therapy, ended therapy to progressive disease, or withdrawn. Low enrollment with most not completing planned therapy, it is not powered for meaningful statistical results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes